CLINICAL TRIAL: NCT03971513
Title: Trans Abdominal Plane Block (TAP Block) in Surgery of Stoma Reversal and Its Effect on Post Operative Recovery: a Prospective, Randomized, Muticenter Study
Acronym: Tapas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RBHP 2019 VIGNAUD - Tapas; 2019-001022-95 (Other: ANSM)
Record Dates: First submitted 2019-05-20; First posted 2019-06-03 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Surgery; Stoma Ileostomy
Keywords: Prospective randomized pilot study; Trans abdominal plane block; Quo R 40 score; Post operative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Model description:
  Randomization in 2 groups
  * Control group (usual practice): patients receiving a general anaesthesia with propofol, sufentanyl and cisatracurium for the induction, and sevoflurane, sufentanyl and cisatracurium for the maintenance. Patients receiving a multimodal intravenous analgesia, with acetaminophen, ketoprophen, nefopam and morphine if necessary Antimicrobial prophylaxis is performed according to recommendations.
  * Experimental group: patients receiving a general anaesthesia with propofol, sufentanyl and cisatracurium for the induction, and sevoflurane, sufentanyl and cisatracurium for the maintenance. Patients receiving a multimodal intravenous analgesia, with acetaminophen, ketoprophen, nefopan and morphine if necessary Antimicrobial prophylaxis is performed according to recommendations. In this group, a trans abdominal plane block, using 20 ml of ropivacaine 5 mg/ml is performed at the beginning of surgery, using ultrasound guidance.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- usual practice (No Intervention): Control group (usual practice): patients receiving a general anaesthesia with propofol, sufentanyl and cisatracurium for the induction, and sevoflurane, sufentanyl and cisatracurium for the maintenance. Patients receiving a multimodal intravenous analgesia, with acetaminophen, ketoprophen, nefopam and morphine. if necessary. Antimicrobial prophylaxis is performed according to recommendations
- TAP block (Experimental): In addition of usual practice, patients receiving a TAP block at the beginning of the surgery
  Interventions: Procedure: Trans abdominal plane

INTERVENTIONS:
Procedure: Trans abdominal plane — Trans abdominal plane block is performed with ultra sound guidance.
  1. - The high frequency probe is placed right to the umbilicus, and slips laterally to the side to block. It allows showing the three belts of larges muscles of abdomen (External Oblicum, internal oblicum, and transversal of the abdomen).
  2. - When the needle is visualised in the plan separating the muscle internal oblicum and transversal of the abdomen, 20 ml of ropivacaïne 5mg/ml are injected after aspiration test. If in doubt, hydro localisation car be realised.
  Arms: TAP block

SUMMARY:
The primary purpose of TAPAS study is to demonstrate the superiority of analgesic effect of trans abdominal plane block (TAP block) performed at the beginning of stoma reversal, compared to standard of care.

The hypothesize is that a TAP block performed at the beginning of surgery of stoma reversal would improve patient's satisfaction (evaluated by Quo-r40 questionnaire), would reduce the incidence of post operative pain, time spent in recovery room, and reduce hospitalisation time

DETAILED DESCRIPTION:
The patient will arrive in the department the day before the surgical intervention (D-1). During this preoperative visit (D-1), the investigator

* will preselect potentially eligible patients
* will offer to participate to this study
* will give the notice form to the patients
* will present the research: objectives, benefits and constraints for the patients

The intervention day (D0):

The investigator will collect the signed consent form after having ascertained the understanding of the notice form by the patient and checking the inclusion and non-inclusion criteria.

The randomization will be done via the eCRF module (allocation group and number) and the preoperative data registration in the eCRF.

Surgical Intervention (D1):

All patients will receive standard anaesthesia using sufentanyl, propopol, cisatracurium and sevoflurane. Prevention of nausea and vomiting is performing using Apfel score. Anti microbial prophylaxis is performed according recommendations.

All patients will receive post operative multimodal analgesia using, acetaminophene, ketaminophene (if no contra indication), nefopam, and morphine if NRS (numerating rating scale) > 3 At the end of the surgery, patients in the experimental group will receive a ultrasound guided trans abdominal plane block with 20 ml of 5 mg/mg of ropivacaine. Patients in the control group will not receive the block

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Patients operated of a scheduled stoma reversal surgery
* Patients having given consent in the mannen described in Article L1122-1-1 of the Public Health Code
* Patients affiliated with asocial security regimen or beneficiary of such a regimen

Exclusion Criteria:

* Renal insufficiency (ie glomerular filtration output < 35 ml/min)
* Patients with chronic inflammatory bowel disease
* Body mass index > 35 kg/m2
* Chronic pain with opiates
* Patients with cognitive troubles
* Coagulation disorders (platelets count < 80G/L, PT< 50%, V factor < 50%)
* Pregnancy
* Breastfeeding
* Local anesthesics (amide class) allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2023-04-17 (Actual)

PRIMARY OUTCOMES:
Quo 40 score | Day 1 (
  Once the patient is transferred in post operative surgical service, assessment of the primary outcome will be done by the physician in charge of the patient. Quo 40 score is a postoperative recovery score above 200 points validated by Myles et al in 2001.

SECONDARY OUTCOMES:
NRS (Numeric rating scale) | Day 1 : At the entrance of recovery room
  Numerating rating score variating from 0 to 10, done by nurses in operating room and in post operative surgical service
NRS (Numeric rating scale) | Day 1
  Numerating rating score variating from 0 to 10, done by nurses in operating room and in post operative surgical service
NRS (Numeric rating scale) | Day 2
  Numerating rating score variating from 0 to 10, done by nurses in operating room and in post operative surgical service
Quo 40 score | Day 15
  Once the patient is transferred in post operative surgical service, assessment of the primary outcome will be done by the physician in charge of the patient. Quo 40 score is a postoperative recovery score above 200 points validated by Myles et al in 2001.
Time spent in recovery room | At the output of recovery room ie until 6 hours after intervention
  Assessment of time spent in recovery room (ie: entrance in recovery room until Aldrede score is >9) performed by nurses (Until 6 hours).

CONTACTS AND LOCATIONS:
Overall Officials: Marie Vignaud, Principal Investigator — CHU Clermont-Ferrand.fr
Locations (2):
- France (2):
  - CHU, Clermont-Ferrand
  - CHU Rennes, Rennes